CLINICAL TRIAL: NCT01152840
Title: Phase II Study of RAD001monotherapy in Patients With Unresectable Adenoid Cystic Carcinoma
Brief Title: Study of RAD001 in Adenoid Cystic Carcinoma
Acronym: ACCRAD001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0710-050-223
Record Dates: First submitted 2010-05-31; First posted 2010-06-29 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2010-06

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: Adenoid cystic carcinoma; RAD001
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Experimental): RAD001 daily po medication
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — RAD001 10 mg po daily medication
  * Treatments will be continued until any of the following events occur:
    * progression of disease,
    * the subject develops unacceptable toxicity,
    * consent to participate in the study is withdrawn.

SUMMARY:
* Although mTOR is clearly an attractive therapeutic target in tumor, no clinical study on mTOR inhibition by RAD001 has been systematically conducted in adenoid cystic carcinoma.
* In phase I study of RAD001, 2 patients with adenoid cystic carcinoma show some response to RAD001 (unpublished data).
* So the investigators design this phase II study of RAD001 in adenoid cystic carcinoma to evaluate the efficacy of RAD001 in this orphan disease.

DETAILED DESCRIPTION:
Although the histologic appearance of adenoid cystic carcinoma is low grade, management of this malignancy is a distinct therapeutic challenge because of its insidious local growth pattern, propensity for perineural involvement, tendency for distant metastasis, and pronounced ability to recur over a prolonged period.

In prospectively performed clinical trials, objective responses to any cytotoxic agent or regimen are infrequent, whereas stabilization of disease was observed more commonly.

In adenoid cystic carcinoma, the study focusing on PI3-K/AKT/mTOR pathway is rare.

According to Younes MN et al's study, adenoid cystic carcinoma cell lines have increased pAkt activity when EGF-stimulation is added. And when treated with EGFR/VEGFR TK dual inhibitor, the phosphorylated form of Akt decreased despite of total level of Akt is remained unchanged.

When the investigators consider that the increased pAkt activity is one of possible predictor to mTOR inhibitor, the mTOR inhibitor might have an activity in adenoid cystic carcinoma.

Although mTOR is clearly an attractive therapeutic target in tumor, no clinical study on mTOR inhibition by RAD001 has been systematically conducted in adenoid cystic carcinoma.

In phase I study of RAD001, 2 patients with adenoid cystic carcinoma show some response to RAD001 (unpublished data).

So the investigators design this phase II study of RAD001 in adenoid cystic carcinoma to evaluate the efficacy of RAD001 in this orphan disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed adenoid cystic carcinoma
* 2. Local, locally-advanced or metastatic disease documented as having shown progression on a scan (CT, MRI, MIBI scan) taken 2 to 12 months prior to baseline compared to a previous scan taken at any time in the past. Progression must be documented according to RECIST criteria.
* 3. Disease that is not amenable to surgery, radiation or combined modality therapy with curative intent and who is previously treated with chemotherapy or local treatment (e,g transarterial chemoembolization)
* 4. Presence of at least one measurable target lesion for further evaluation according to RECIST criteria
* 5. 18 years or older
* 6. ECOG performance status 0, 1
* 7. Previous treatment with chemotherapy, loco-regional therapy (e.g chemoembolization) are permitted providing that toxicity has resolved to ≤grade 1 at study entry and that last treatment was at least 4 weeks prior to baseline assessment.
* 8. Adequate organ function
* 9. A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
* 10. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

* 1. A patient with no measurable disease
* 2. Prior chemotherapy, radiation therapy or surgery within 4 weeks prior to study entry except palliative radiotherapy to non-target lesions (within 2 weeks prior to study entry)
* 3. A patient with previous active or passive immunotherapy
* 4. A patient with intestinal obstruction or impending obstruction, recent active upper GI bleeding
* 5. A pregnant or lactating patient
* 6. A patient of childbearing potential without being tested for pregnancy at baseline or with being tested for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential)
* 7. A man or woman of childbearing potential who has no willingness to use a contraceptive measure during the study
* 8. A patient with history of another malignant disease within past 5 years, except curatively treated basal cell carcinoma of skin and cervical carcinoma in situ.
* 9. A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.
* 10. A patient with clinically significant heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmia, etc) or myocardial infarction within past 12 months.
* 11. Ongoing cardiac arrhythmia of grade ≥2, atrial fibrillation of any grade, or QTc interval>450msec for males or >470msec for female.
* 12. A patient with interstitial pneumonia or diffuse symptomatic fibrosis of the lungs
* 13. A patient with peripheral neuropathy of grade 1 by NCI CTC, caused by other factors (e.g. alcohol, diabetes, etc). If the absence of deep tendon reflexes is the only neurologic disorder, this condition does not apply to the exclusion criteria.
* 14. A patient with organ transplantation requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
progression free survival rate at 4 months | 10 months
  proportion of patients who are alive and progression-free at the time of 4 months of treatment among all patients

SECONDARY OUTCOMES:
the time to progression (TTP) | 10 months
overall survival (OS) | 2 years
response rate (RR) | 6 months
the metabolic response rate by PET-CT | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, MD, PhD, Principal Investigator — Seoul National University Hospital; Do-Youn Oh, MD,PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim DW, Oh DY, Shin SH, Kang JH, Cho BC, Chung JS, Kim H, Park KU, Kwon JH, Han JY, Kim MJ, Bang YJ. A multicenter phase II study of everolimus in patients with progressive unresectable adenoid cystic carcinoma. BMC Cancer. 2014 Nov 3;14:795. doi: 10.1186/1471-2407-14-795. PMID 25362970